CLINICAL TRIAL: NCT00119002
Title: The Effectiveness of Oral Dexamethasone for Acute Bronchiolitis: A Multicenter Randomized Controlled Trial
Brief Title: The Effectiveness of Oral Dexamethasone for Acute Bronchiolitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Children's Hospital of Michigan (Other); Children's Hospital Medical Center, Cincinnati (Other); Washington University School of Medicine (Other); Columbia University (Other); Children's National Research Institute (Other); Helen DeVos Children's Hospital (Other); Women & Children's Hospital of Buffalo (Other); University of Rochester (Other); NYU Langone Health (Other); Hurley Medical Center (Other); Boston Children's Hospital (Other); University of Maryland (Other); Johns Hopkins University (Other); Howard County General Hospital (Unknown); University of California, Davis (Other)
Responsible Party: Howard Corneli, MD Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R40MC04298-01-00
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-01

CONDITIONS: Bronchiolitis, Viral
Keywords: randomized clinical trial; placebo-controlled; double-blind; double-masked; infant; dexamethasone; wheezing
MeSH Terms: conditions — Bronchiolitis, Viral; Respiratory Sounds | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Active Comparator): 1mg of Dexamethasone/kg
  Interventions: Drug: dexamethasone
- Placebo (Placebo Comparator): 1mg/kg placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dexamethasone — 1mg/kg dexamethasone
  Arms: Dexamethasone
Drug: Placebo — 1mg/kg placebo
  Arms: Placebo

SUMMARY:
This study will compare a single dose of oral dexamethasone to placebo in a multicenter, randomized, double blind trial of infants aged 2 to 12 months with first-time bronchiolitis (defined as wheezing within 7 days of onset). This is given as additional therapy beyond any other routine therapy used at that center. No current standard therapy is withheld, and no additional tests or other treatments are part of the study.The primary hypothesis is that dexamethasone will be more effective than placebo in preventing hospital admission. The secondary hypotheses are that dexamethasone will decrease respiratory scores and possibly the duration of the disease when compared to placebo, and that dexamethasone will be as safe and as well tolerated as placebo.

DETAILED DESCRIPTION:
Bronchiolitis is the most common lower respiratory infection in infants, and the respiratory condition leading to the most hospital admissions in young children. It is also probably the most common serious illness of childhood lacking evidence-based treatment. Evidence both for and against the effectiveness of corticosteroids such as dexamethasone has been published. Editorials, expert reviews, and a recent report from the Agency for Healthcare Research and Quality recommend a study such as this one.

Patients will be drawn from the emergency departments at participating medical centers in the Pediatric Emergency Care Applied Research Network, created by the Emergency Medical Services for Children program and the Maternal and Child Health Bureau of the Health Resources and Services Administration to study health problems of high acuity and high incidence in children.

Comparisons: The primary outcome (hospital admission after 4 hours of ED observation) and secondary outcomes will be compared between treatment and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* First attack of wheezing within 7 days of onset
* Age 2 months through 11 months (less than 12 months)
* Disease of at least moderate severity (RDAI score greater than or equal to 6)

Exclusion Criteria:

* Prior adverse reaction to dexamethasone
* Known heart or lung disease
* Premature birth prior to 36 weeks' gestation
* History of prior asthma or bronchodilator use
* Immune suppression or deficiency
* Trisomy 21
* Critical or life-threatening complications of bronchiolitis
* Treatment with corticosteroids within 14 days
* Known active chickenpox
* Exposure to chickenpox within 21 days
* Child sent to ED for automatic admission

Ages: 2 Months to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 598 (Actual)
Dates: Start 2004-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Hospital admission after 4 hours of ED observation | 4 hours

SECONDARY OUTCOMES:
Severity of disease measured by respiratory (RDAI) scores, vital signs, and oximetry. | 4 hours
Duration of hospitalization (if admitted) measured at 7-to-10 day followup. | 7-10 days
Safety, toleration, and parental satisfaction measured at 7-to-10 day followup. | 7-10 days

CONTACTS AND LOCATIONS:
Overall Officials: Howard Corneli, MD, Principal Investigator — University of Utah
Locations (1):
- Primary Children's Medical Center, Salt Lake City, Utah, United States

REFERENCES:
- [Result] Corneli HM, Zorc JJ, Mahajan P, Shaw KN, Holubkov R, Reeves SD, Ruddy RM, Malik B, Nelson KA, Bregstein JS, Brown KM, Denenberg MN, Lillis KA, Cimpello LB, Tsung JW, Borgialli DA, Baskin MN, Teshome G, Goldstein MA, Monroe D, Dean JM, Kuppermann N; Bronchiolitis Study Group of the Pediatric Emergency Care Applied Research Network (PECARN). A multicenter, randomized, controlled trial of dexamethasone for bronchiolitis. N Engl J Med. 2007 Jul 26;357(4):331-9. doi: 10.1056/NEJMoa071255. PMID 17652648
- See also: Pediatric Emergency Care Applied Research Network (PECARN) — http://www.pecarn.org